CLINICAL TRIAL: NCT02975765
Title: Evaluation of the Levels of Pain and Discomfort Between Piezosurgery-assisted Corticotomy Versus Traditional Method of Aligning Crowded Lower Anterior Teeth: a Randomized Controlled Trial
Brief Title: Evaluation of the Levels of Pain and Discomfort Between Two Methods of Correcting Misaligned Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OMFS-02-2016
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Malocclusion; Crowded Teeth; Surgical Incision
Keywords: corticotomy; minimally invasive; piezosurgery; piezocision; pain; discomfort
MeSH Terms: conditions — Malocclusion; Crowding; Surgical Wound; Pain | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Piezosurgery (Experimental): Piezosurgery-assisted corticotomy will be performed to enhance teeth alignment
  Interventions: Procedure: Piezosurgery
- Traditional method (No Intervention): No intervention is going to be applied to the patients in this group.

INTERVENTIONS:
Procedure: Piezosurgery — The surgical tip is going to be used to make small cuts into the cortex of the alveolar bone between the crowded teeth.
  Other Names: Piezocision
  Arms: Piezosurgery

SUMMARY:
Applying flapless piezocision corticotomies on the alveolar bone and separating anterior mandibular teeth using a piezosurgery device (i.e. ultrasonic waves that perform very accurate incisions without any sutures following this procedure) may improve the speed of tooth alignment during orthodontic treatment. This study consists of two groups, patients will be randomly assigned to one of these two groups. The levels of pain and discomfort of this procedure on 18 patients (experimental group) will be evaluated,whereas the second group (control group) will receive a traditional orthodontic therapy.

DETAILED DESCRIPTION:
According to the American Association of Orthodontists (AAO), the length of comprehensive orthodontic treatment ranges between 18-30 months, depending on treatment options and individual characteristics. In addition, orthodontic treatment time ranges between 25-35 months for extraction therapies, respectively. Reducing orthodontic treatment time is one of the main goals for orthodontists, due to problems such as root resorption, periodontal disease and caries that are associated with prolonged treatment time.

Many techniques have been introduced to accelerate orthodontic tooth movement; surgical and non-surgical. The surgical approach is the most clinically applied and most tested with known predictions and stable results. Surgical approaches usually vary from total block osteotomies to flapless partial corticotomies .In spite of corticotomy-assisted orthodontic treatment efficiency, the invasiveness of these procedures (i.e. requiring full mucoperiosteal flaps elevation) might have limited their widespread acceptance among orthodontists and patients. Therefore, more conservative flapless corticotomy techniques have recently been proposed. These procedures can be accomplished in a reasonably short periods that might produce less pain and discomfort, so we will gain better patient acceptance. Although various techniques of flapless corticotomy have been reported to be successful in practice, scientific evidence on their acceptance and compatibility is little in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients , Male and female, Age range: 16-26 years.
2. Severe crowding ≤ 7 (Little's irregularity index)
3. Permanent occlusion.
4. Exist all the Mandibular teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth<4 mm
   * No radiographic evidence of bone loss .
   * Gingival index≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, NSAIDs, …)
2. Patients have anti indication for oral surgery ( medical - social - psycho)
3. Presence of primary teeth in the mandibular arch
4. Missing permanent mandibular teeth (except third molars).
5. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
6. Patient had previous orthodontic treatment

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12-12 (Actual); Study Completion 2017-04-23 (Actual)

PRIMARY OUTCOMES:
Levels of Pain and Discomfort at one day | at 24 hours following the engagement of first initial arch wire in the brackets
  Pain and discomfort will be measured on visual analog scale
Levels of Pain and Discomfort at seven days | at seven days following the onset of orthodontic treatment
  Pain and discomfort will be measured on visual analog scale
Levels of Pain and Discomfort at 14 days | at 14 days following the onset of orthodontic treatment
  Pain and discomfort will be measured on visual analog scale
Levels of Pain and Discomfort at 28 days | at 28 days following the onset of orthodontic treatment
  Pain and discomfort will be measured on visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Omar Gibreal, DDS, Principal Investigator — MSc student, Oral and Maxillofacial Surgery Department, University of Damascus Dental School; Bassel Brad, DDS MSc PhD, Study Director — Associate Professor of Oral and Maxillofacial Surgery, Department of Oral and Maxillofacial Surgery, Univ. of Damascus Dental School; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, Department of Orthodontics, University of Damascus Dental School
Locations (1):
- Departments of Orthodontics and Oral and Maxillofcial Surgery, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sebaoun JD, Surmenian J, Dibart S. [Accelerated orthodontic treatment with piezocision: a mini-invasive alternative to conventional corticotomies]. Orthod Fr. 2011 Dec;82(4):311-9. doi: 10.1051/orthodfr/2011142. Epub 2011 Nov 23. French. PMID 22105680
- [Background] Vercellotti T, Podesta A. Orthodontic microsurgery: a new surgically guided technique for dental movement. Int J Periodontics Restorative Dent. 2007 Aug;27(4):325-31. PMID 17726988
- [Background] Keser EI, Dibart S. Sequential piezocision: a novel approach to accelerated orthodontic treatment. Am J Orthod Dentofacial Orthop. 2013 Dec;144(6):879-89. doi: 10.1016/j.ajodo.2012.12.014. PMID 24286911
- [Derived] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984